CLINICAL TRIAL: NCT04616911
Title: External Anal Sphincter-Sparing Seton After Rerouting Versus Ligation of Intersphincteric Fistula Tract (LIFT) In Treatment Of Complex Anal Fistula: A Randomized Clinical Trial
Brief Title: Rerouting Seton Versus LIFT for Complex Anal Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Associate professor of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mansoura2020M
Record Dates: First submitted 2020-11-01; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rerouting seton (Active Comparator): Placement of seton with rerouting of the fistula tract around the internal anal sphincter
  Interventions: Procedure: Rerouting seton
- LIFT (Active Comparator): Ligation of the intersphincteric fistula tract
  Interventions: Procedure: LIFT

INTERVENTIONS:
Procedure: Rerouting seton — Excision of superficial fistula tract and placment of seton with rerouting of the fistula tract around the internal anal sphincter
  Arms: Rerouting seton
Procedure: LIFT — Ligation of the intersphincteric fistula tract
  Arms: LIFT

SUMMARY:
This study aims to compare the efﬁcacy of two surgical techniques in treatment of complex anal fistulas. The first technique involves rerouting of the fistula tract with placement of a vessel loop seton around the internal anal sphincter, sparing the external sphincter whereas the second technique entails ligation of inter-sphincteric fistulous tract (LIFT). The main objectives of the study are to assess the success rate, time to healing, change in quality of life, and complications of each procedure including fecal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex with complex anal fistula including high trans-sphincteric, supra-sphincteric, extra-sphincteric, and anterior fistula in female

Exclusion Criteria:

* Patients with simple anal fistulas, including intersphicnteric and low trans-sphincteric fistulas.
* ASA IV and V (The American Society of Anesthesiologists Physical Status classification system) unfit patients
* Patient with any grade of anal incontinence.
* Patients with concomitant anal pathology.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Healing of anal fistula | 12 months after surgery
  Clinical healing is assessed by clinical examination during follow-up and is defined as Complete epithelization of the anal wound with no residual fistula tract or external opening or discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., FACS, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No